CLINICAL TRIAL: NCT05904782
Title: Development of Brief Positive Affect Treatment (PAT) for Caregivers of Patients With Advanced Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0940; NCI-2023-04226 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To learn more about the experience and wellbeing of people who provide care for cancer patients.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objectives:

The primary objective of this proposal is to identify relevant themes and content essential to adapt PAT to a caregiving in advanced cancer context (PAT-C) and develop a Brief (5-session) version of PAT-C. Findings from this study are essential to inform future RCTs to test the feasibility, efficacy, dose and explore potential mediators of treatment outcomes of this intervention.

Secondary Objectives:

The secondary objective is to characterize psychosocial distress and psychosocial health of caregivers in the supportive care clinic. This data will be essential to inform appropriateness of the supportive care clinic as a potential site for future RCTs (i.e., determine if there are enough caregivers in this clinic who might benefit from this specific supportive care strategy).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Males and female adults ≥18 years
* Able to read and speak English
* Caregiver of a patient diagnosed with stage IV solid malignancy, with whom they have been residing for >6 months
* Access to necessary resources for participating in a technology-based intervention (i.e., telephone, internet access)

Exclusion Criteria:

* Current participation in consistent (self-defined) psychotherapy
* Caregivers who are considered part of a vulnerable population (i.e. cognitively impaired (self-reported or patient-reported), pregnant, military personnel) will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life questionnaire (Qol) | through completion of study; approximately 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Kroll, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org